CLINICAL TRIAL: NCT01246310
Title: Myoinositol for the Treatment of Ovarian and Psychiatric Disorder in PCOS Patients.
Brief Title: Myoinositol for the Treatment of Ovarian and Psychiatric Disorder in Polycystic Ovary Syndrome (PCOS) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of patients enrolled was insufficient to match the calculated sample size and to carry out statistical analyses
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Collaborators: Centro Clinico Colle Cesarano Tivoli Rome Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: agunco7/2010
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Depression; PCOS
MeSH Terms: conditions — Depression | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inositol (Experimental)
  Interventions: Dietary Supplement: Inositol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inositol
  Arms: Inositol
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common reproductive disorders affecting 5-10% of women of reproductive age. Beside impairments on reproductive functions (oligomenorrhea/amenorrhea), it also affects metabolism (insulin resistance, type 2 diabetes mellitus and cardiovascular risk) and psychology (increased anxiety, depression and eating disorders). Recently, several studies have shown that there is an increased risk of mood disorders in women with PCOS, with major depression and bipolar disorder as the most frequent diagnosis.

Myo-inositol is classified as a member of the vitamin B complex and it works as a second messenger system of several neurotransmitter receptors; furthermore, inositol, when administrated at pharmacological doses, crosses the blood-brain barrier.

Studies from the 90s showed that inositol, alone or in combination with other antidepressant drugs (mainly serotonin reuptake inhibitors), is able to induce improvement of the Hamilton depression rating Scale.

Recently, inositol has been proposed as treatment to improve clinical, metabolic and endocrinal status in PCOS patients. Administration of myo-inositol to PCOs patients resulted in several beneficial effects, such as decrease of circulating insulin and serum total testosterone as well as a restored ovulation.

In this proposed study, the investigators aim to evaluate in a double blind randomized trial whether inositol alone has beneficial effects on mental health disorders associated with PCOs. In particular, 60 women in reproductive age that will be diagnosed of PCOs, according to Rotterdam 2003 criteria, will be recruited and randomly assigned to the inositol or placebo group. Both groups will go through ultrasonic evaluation of the ovaries and serum hormonal levels (FSH, LH, testosterone, estradiol and insulin) will be evaluated. Furthermore, with the help of psychiatrics, patients will be interviewed in order to test the presence of any mental health disorders using validated tests such as: Hamilton Anxiety Scale (HAM-A), Hamilton Rating Scale for Depression (HAM-D), Health Assessment Questionnaire (HAQ), Short Form of Mc Gill Pain Questionnaire (SF-MPQ).

Women assigned to the inositol group will receive 12g of inositol during the day in three different administrations for a period of 4weeks.

At the end of treatment period patients will be interviewed by psychiatrics and will go through ultrasonic evaluation of the ovaries and hormonal levels will be tested

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed of PCOS according to Rotterdam 2003 criteria

Exclusion Criteria:

* BMI >30
* Pharmacological treatment in the last 3 moths
* Use of contraceptive pill

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for depression
Hamilton Anxiety Scale
Health assessment Questionnaire
Short form of Mc Gill Pain Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Unfer, MD, Principal Investigator — AGUNCO Obstetrics and Gynecology Centre; Buffo Silvia, MD, Principal Investigator — Centro Clinico Colle Cesarano Tivoli Rome Italy
Locations (1):
- Agunco, Rome, Italy

REFERENCES:
- [Background] Costantino D, Minozzi G, Minozzi E, Guaraldi C. Metabolic and hormonal effects of myo-inositol in women with polycystic ovary syndrome: a double-blind trial. Eur Rev Med Pharmacol Sci. 2009 Mar-Apr;13(2):105-10. PMID 19499845
- [Background] Levine J, Barak Y, Gonzalves M, Szor H, Elizur A, Kofman O, Belmaker RH. Double-blind, controlled trial of inositol treatment of depression. Am J Psychiatry. 1995 May;152(5):792-4. doi: 10.1176/ajp.152.5.792. PMID 7726322
- [Background] Kerchner A, Lester W, Stuart SP, Dokras A. Risk of depression and other mental health disorders in women with polycystic ovary syndrome: a longitudinal study. Fertil Steril. 2009 Jan;91(1):207-12. doi: 10.1016/j.fertnstert.2007.11.022. Epub 2008 Feb 4. PMID 18249398
- [Background] Papaleo E, Unfer V, Baillargeon JP, Chiu TT. Contribution of myo-inositol to reproduction. Eur J Obstet Gynecol Reprod Biol. 2009 Dec;147(2):120-3. doi: 10.1016/j.ejogrb.2009.09.008. Epub 2009 Oct 2. PMID 19800728
- [Background] Teede H, Deeks A, Moran L. Polycystic ovary syndrome: a complex condition with psychological, reproductive and metabolic manifestations that impacts on health across the lifespan. BMC Med. 2010 Jun 30;8:41. doi: 10.1186/1741-7015-8-41. PMID 20591140
- [Background] Baptiste CG, Battista MC, Trottier A, Baillargeon JP. Insulin and hyperandrogenism in women with polycystic ovary syndrome. J Steroid Biochem Mol Biol. 2010 Oct;122(1-3):42-52. doi: 10.1016/j.jsbmb.2009.12.010. Epub 2009 Dec 28. PMID 20036327